CLINICAL TRIAL: NCT02246205
Title: Billroth II or Roux-en-Y Reconstruction for Gastrojejunostomy After Pancreaticoduodenectomy: Randomized Controlled Trial (PAUDA TRIAL): Comparison of Morbidity and Delayed Gastric Emptying
Brief Title: Billroth II or Roux-en-Y Reconstruction for GJ After PD: Randomized Controlled Trial (PAUDA TRIAL)
Acronym: PAUDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, JULI BUSQUETS BARENYS, Medicine Doctor, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAUDA
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Malignant Neoplasm of Head of Pancreas
Keywords: pancreaticoduodenectomy; delayed gastric emptying; Roux en-Y reconstruction
MeSH Terms: conditions — Gastroparesis | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DPC DN (Experimental): Roux-en Y reconstruction after pancreaticoduodenectomy
  Interventions: Procedure: Pancreaticoduodenectomy
- DPC UN (Active Comparator): Child reconstruction after pancreaticoduodenectomy
  Interventions: Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy — Pancreaticoduodenectomy is the classical operative technique to resect cephalic pancreatic cancer. In a first phase of the surgery, the resection may be performed. In the second phase, the digestive tract must be restored. We planify two different reconstruction techniques.

SUMMARY:
The aim of the study is to compare the effect of Roux-en Y reconstruction (study group, DPCDA) versus classical Child reconstruction (DPCUN) in the incidence of VGL in patients for DPC. The hypotesis of the study is that Roux-en Y reconstruction decreases incidence of DGE after pancreaticoduodenectomy.

DETAILED DESCRIPTION:
The pancreaticoduodenectomy (DPC) is the procedure of choice of the tumors of the head of the pancreas, periampullary tumors and intractable inflammatory pathology.

The high postoperative morbidity (50%) involve a mean hospital stay of 15 days after surgery. The most common complication is delayed gastric emptying (DGE), defined as the intolerance to solid oral intake by 7th day postoperative. In some severe cases, oral intolerance can occur after the 21th postoperative day. Therefore, the patient requires parenteral nutrition and prolonged hospital stay.

The aim of the study is to compare the effect of Roux-en Y reconstruction (study group, DPCDA) versus classical Child reconstruction (DPCUN) in the incidence of VGL in patients for DPC.

The hypotesis of the study is that Roux-en Y reconstruction decreases incidence of DGE after pancreaticoduodenectomy.

A pilot randomized clinical trial has been designed to compare two surgical techniques for reconstruction of digestive tract after DPC in patients treated in our center. The patients are randomized after tumor resection and before the reconstruction througt computer-generated random numbers using a sealed envelope technique. The primary endpoint is the incidence of DGE. Secondary endpoints are postoperative morbidity and specific complications as pancreatic fistula, the hospital stay, and postoperative endocrine and exocrine function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic head cancer considered resectable after the extension study
* Patients suffering from periampullary tumors considered resectable after the extension study
* Patients suffering from pancreatic inflammatory disease with medically intractable pain
* Patients who have read the information sheet of the study and signed the informed consent form

Exclusion Criteria:

* Patients with history of previous gastrectomy
* Patients with associated resections of other organs, except for the superior portal vein or mesenteric vein
* Patients with enlargement to total pancreatectomy
* Patients who has recieved neoadjuvant treatment
* Patients with plastic peritonitis
* Patients with liver cirrhosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Delayed gastric emptying incidence after pancreaticoduodenectomy | within the first 60 daysafter surgery
  DGE, defined as oral diet intolerance from the 7th postoperative day, and the persistence of nasogastric tube on the 4th postoperative day or later, according to the ISGPS criteria

SECONDARY OUTCOMES:
Morbidity and complications after pancreaticoduodenectomy | within the first 60 daysafter surgery
  Postoperative morbidity was defined as any complication that appeared during hospital admission. Postoperative complications and postoperative mortality were defined according to the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: JULI BUSQUETS, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, Hospitalet Llobregat, Barcelona, Spain